CLINICAL TRIAL: NCT05822297
Title: Myokines and Cognitive Aging in People With Spinal Cord Injury: a Single Case Experimental Design Study
Brief Title: SCED Myokines and Cognition in SCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Adelante, Centre of Expertise in Rehabilitation and Audiology (Other)
Responsible Party: Principal Investigator, Wouter Vints, Principal Investigator, Adelante, Centre of Expertise in Rehabilitation and Audiology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CoBes22.055
Record Dates: First submitted 2023-04-07; First posted 2023-04-20 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-12

CONDITIONS: Spinal Cord Injuries; Cognitive Decline
Keywords: Aging; Myokine; Cognition; Spinal cord injury; Neuromuscular electrical stimulation
MeSH Terms: conditions — Spinal Cord Injuries; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: A single case experimental design (SCED) with sequential multiple baseline time series and a single-armed prospective study design, with a random duration of the baseline phase ranging from 3 to 6 weeks, an intervention phase of 12 weeks, and a 12 week period without measurements, followed by a follow-up phase of 3 weeks; in addition to a single-armed prospective study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): Each participant will undergo the same procedures and intervention, consisting of a baseline phase, intervention phase and follow-up phase. The length of the baseline phase will be randomized 3, 4, 5 or 6 weeks.
  Interventions: Device: Neuromuscular electrical stimulation

INTERVENTIONS:
Device: Neuromuscular electrical stimulation — NMES will consist of a 12 week electrical stimulation program, three times a week. Electrical stimulation will be done on the quadriceps muscles of both legs simultaneously. For each leg, one electrode is placed on the proximal side and one on the distal side of the quadriceps muscle. Electrical stimulation sessions will take 30min, at a stimulation frequency of 50Hz, an intensity where we can at least see a visible or palpable contraction with a maximum intensity of 100mA (we will choose the highest intensity that is easily supported by the participant without inducing discomfort) and a pulse width of 400μs. The activation within the activation-rest cycle consists of a 1s ramp-up, 7s full activation and 1s ramp-down, followed by 18s rest. Every 4 weeks the rest period will be diminished with 3s until a total of 9s.

SUMMARY:
Rationale: Individuals with spinal cord injury (SCI) suffer from accelerated cognitive aging. In able-bodied individuals, a vast amount of studies have shown that exercise interventions can improve cognitive function. Myokines (i.e. factors released into the blood stream from muscle cells) are considered one of the mediators of this beneficial effect. Neuromuscular electrical stimulation (NMES), used to replace or support muscle training in disabled individuals with poor exercise possibilities, was shown to elicit a large release of myokines (in some studies larger than following voluntary exercise). However, so far, the effects of NMES on cognitive function have never been studied before. In fact, only one study has previously investigated the effect of exercise on cognitive function in persons with SCI.

Objective: The primary aim is to assess to what extent a 12 week intervention with NMES to the quadriceps muscles of people with SCI can change their performance on a set of cognitive tests. Secondarily, the investigators will measure to what extent NMES to the quadriceps muscles of people with SCI induces changes in blood levels of the myokine brain-derived neurotrophic factor (BDNF), which is considered a potential mediator of the exercise-cognition effect, facilitating neuroplastic processes.

Study design: A single case experimental design (SCED) with sequential multiple baseline time series and a single-armed prospective study design, with a random duration of the baseline phase ranging from 3 to 6 weeks, an intervention phase of 12 weeks, and a 12 week period without measurements, followed by a follow-up phase of 3 weeks; in addition to a single-armed prospective study design.

Study population: Individuals (n = 15) aged 18 years and older with a chronic SCI (>1y post-injury) and with visible or palpable contraction of the quadriceps muscles upon NMES will be recruited at the rehabilitation centre of Adelante in Hoensbroek, the Netherlands.

Intervention: The study participants will receive 30min of NMES using surface electrodes on the quadriceps muscles three times per week for a total duration of 12 weeks.

Main study parameters/endpoints: The primary outcome is cognitive function changes which will be measured using a secured smartphone application (e.g. m-Path). Secondary outcome measures are changes in the blood myokine levels of BDNF and changes in cognitive outcome scores on an verbal cognitive test battery.

ELIGIBILITY:
Inclusion Criteria:

* Persons with spinal cord injury
* Completeness of injury: American Spinal Injury Association (ASIA) Impairment Scale (AIS) A, B or C
* Level of injury: L2 or higher
* At least 18 years old
* Chronic stage (> 1 year) since injury
* No previous surgery to the quadriceps muscles
* Intact hand function
* Able to use apps on smartphone (i.e. participants should have their own smartphone and should not have disabilities that impair them to operate it independently)
* Able to follow the instructions of placing the surface electrodes of the NMES device correctly or to have someone else put the electrodes for them
* Dutch as a native language

Exclusion Criteria:

* Malignant processes, or history of undergoing chemotherapy, or history of radiotherapy to the head
* No visible or palpable contraction of the quadriceps muscle upon electrical stimulation
* Intolerance to electrical stimulation of the quadriceps muscle
* Recent or current participation in an electrical stimulation-induced exercise or therapy program in which regular electrical stimulation was given (up to 6 months prior to study inclusion)
* Known neurodegenerative disorder, such as Alzheimer's disease or Parkinson's disease
* Known psychiatric disorder, such as major depressive disorder or bipolar disorder
* Current pressure ulcer
* History of severe autonomic dysreflexia
* Metal implants in the electrical stimulation area
* Intrathecal baclofen (ITB) device
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Change in executive function | measured a total of 54-63 times in 30-33 weeks time
  response time (in ms) on the momentary digital symbol substitution task

SECONDARY OUTCOMES:
Neurocognitive test battery, change in cognitive scores | before and after the 12 week intervention and after a 12 week follow-up
  A neurocognitive test battery will be used to assess cognitive changes on various cognitive domains over time
Concentration of brain-derived neurotrophic factor (BDNF) | before and after the 12 week intervention and after a 12 week follow-up
  Brain-derived neurotrophic factor will be measured in blood of the participants
Self-perceived cognitive function | before and after the 12 week intervention and after a 12 week follow-up
  measured using the cognitive failures index (CFI), ranging from 0-100, with a higher score indicating more subjective cognitive problems
Pain score | before and after the 12 week intervention and after a 12 week follow-up
  measured using the McGill Pain Questionnaire (MPQ), ranging from 0-78, with a higher score indicating higher subjective pain level
Fatigue | before and after the 12 week intervention and after a 12 week follow-up
  measured using the Fatigue Severity Scale (FSS), ranging from 1-7, with a higher score indicating more fatigue/higher impact of fatigue on daily activities
Participation in daily life activities | before and after the 12 week intervention and after a 12 week follow-up
  measured using the Utrecht Scale for Evaluation of Rehabilitation-Participation (USER-P), ranging from 0-100, with a higher score indicating larger participation in daily life activities
Spasticity | before and after the 12 week intervention
  measured using the Perceived Resistance to Passive Movement (PRPM) test at all four limbs.
Electrically-evoked quadriceps strength | before and after the 12 week intervention
  measured using the MicroFET2 dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte van Laake, MD, PhD, Principal Investigator — Center of Exertise in Rehabilitation and Audiology, Adelante Zorggroep
Locations (1):
- Adelante Zorggroep, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No
All information will be coded and kept behind locked doors.

REFERENCES:
- [Derived] Vints WAJ, Levin O, van Griensven M, Vlaeyen JWS, Masiulis N, Verbunt J, van Laake-Geelen CCM. Neuromuscular electrical stimulation to combat cognitive aging in people with spinal cord injury: protocol for a single case experimental design study. BMC Neurol. 2024 Jun 11;24(1):197. doi: 10.1186/s12883-024-03699-9. PMID 38862912